CLINICAL TRIAL: NCT04327102
Title: Health Management Model Construction and Effect Evaluation of Hypertension Patients Based on Disease-related Health Literacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huzhou Normal University (Other)
Responsible Party: Principal Investigator, ZHANG Qing-hua, Associate Professor, Ph.D, Huzhou Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HuzhouNormalU
Record Dates: First submitted 2020-02-29; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Health Literacy; Hypertension
Keywords: health literacy; hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental : intervention group (Experimental): Combination of health education tools and health literacy intervention: on the basis of the control group, the hypertension health education tools are used as the education media to encourage patients to find out the elements of the tool chart, use the picture content to guide the topic development, encourage patients to discuss with each other, realize heuristic questions, rather than a single indoctrination, so as to deepen the understanding and memory of patients. At the end of the course, patients are encouraged to set short-term goals to encourage behaviors that continue to achieve larger goals. At the same time, health literacy lectures were organized during the hospitalization. Health literacy lecture is mainly to learn the information that hypertension needs to pay attention to in order to improve the health literacy of hypertension patients and other indicators.
  Interventions: Behavioral: Health education tools combined with health literacy intervention
- No intervention:The control group (No Intervention): No intervention except conventional care were performed for the control group

INTERVENTIONS:
Behavioral: Health education tools combined with health literacy intervention — On the basis of the control group, the intervention measures to improve the health literacy of patients were implemented and self-made health education tools were used. During hospitalization, health knowledge lectures shall be organized for patients. Before the activity, the theme of the activity shall be clarified. Each participant shall be organized by the educator to sit on the tool chart in a U-shape. According to the theme of the tool map, patients interact with educators. And learn the knowledge content related to hypertension health literacy. Before the end of the activity, the educator will review all the contents discussed in the activity quickly, answer the questions in the activity, and help the participants to sort out and consolidate the knowledge acquired in the education. Follow up intervention for patients after leave hospital.
  Arms: Experimental : intervention group

SUMMARY:
Huzhou City, Zhejiang Province was chosen as the research site, and a general hospital was randomly selected. The "Chinese version of hypertension health literacy scale" of the tutor of this research group was used to evaluate the health literacy level of inpatients with hypertension in the Department of Cardiology, and the patients with critical and lack of health literacy were selected as the research objects. In the control group, routine health management was carried out. On the basis of the control group, the intervention group used health education tools combined with health literacy intervention to implement interactive health management for 12 months. The results of the intervention measures were compared to evaluate the effects of the intervention measures on improving the health literacy level, Hypertension Self-care ability, quality of life and reducing systolic and diastolic blood pressure, body mass index, waist circumference, physiological and biochemical indicators of the patients, so as to provide theoretical basis and practical reference for the further development of prevention and treatment strategies of hypertension patients.

DETAILED DESCRIPTION:
First, the Chinese version of hypertension health literacy scale was used to evaluate the health literacy of inpatients in a hospital, and then the critical and lack of health literacy patients were selected as the research objects.

Then, taking a place in Huzhou City of Zhejiang Province as the research site, a general hospital was randomly selected. According to the ratio of male to female = 1:1, the hypertension patients who meet the inclusion criteria were screened until the intervention group and the control group reached the required sample size. Patients were randomly assigned to the intervention group and the control group.

After the patients signed the informed consent, the patients were intervened. Finally, data collection and statistical processing are carried out

ELIGIBILITY:
Inclusion Criteria：

* Age ≥ 16 years old and has lived in Huzhou for nearly half a year;
* The Chinese version of the hypertension health literacy scale was used to evaluate the health literacy of those with a total score of less than 32 + the critical group;
* In line with the diagnostic criteria for essential hypertension set out in China's hypertension prevention and control guidelines in 2018, systolic blood pressure ≥ 140mmHg, and / or diastolic blood pressure ≥ 90mmHg;
* In the last half year, the living condition is stable, and there is no major stress event (such as the death of relatives, etc.);
* Volunteer to participate in the study, and sign the informed consent of research willingness.

Inclusion Criteria：

* All kinds of secondary hypertension patients;
* Major stress events occurred during the study period;
* Have serious mental disorder or serious cognitive function defect;
* Patients with severe acute and chronic physical diseases；
* Cardiovascular risk factors: low risk or high risk.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
High Blood Pressure-Health Literacy Scale into Chinese | 12 months
  The scale consists of 15 items and 5 dimensions, with a total score of 0-60. One score will be given if one question is answered correctly. The higher the score is, the higher the HL level is. According to the TOFHLA classification standard, HL level is divided into three levels. If the score is less than 32, the HL level is deficient; if the score is 32-40, the HL level is critical; if the score is more than 40, the HL level is sufficient. The score of the scale before and after the intervention was compared.
Systolic and diastolic blood pressure in hypertension | 12 months
  The decrease of systolic and diastolic blood pressure in hypertension patients after health literacy intervention
Body Mass Index ，BMI | 12 months
  According to 2008 WHO guidelines, BMI < 25 kg / m2 is normal weight or low weight, 30 kg / m2 > BMI ≥ 25 kg / m2 is overweight, BMI ≥ 30 kg / m2 is obesity. To evaluate the changes of BMI of patients before and after intervention
Waist Circumference，WC | 12 months
  WC ≥ 102CM in male and 88cm in female were abdominal obesity, 94cm ≤ male WC < 102CM, 80cm ≤ female WC < 88cm are abdominal overweight, WC < 94cm in male and 80cm in female is normal.To evaluate the changes of WC of patients before and after intervention
Quality of Life Instruments for Chronic Diseases - Hypertension V2.0: scale scores | 12 months
  The scale consists of 41 items and uses the five point equidistant scoring method. The scores are 1, 2, 3, 4 and 5 in turn. The total score of the scale is between 41 and 205. The higher the score, the better the quality of life.Compare the changes of the scale scores before and after the intervention
Chinese version of Hypertension Self-care Profile | 12 months
  There are 60 items in the scale. Each item in the scale is 1-4 points, and the total score of the scale is 60-240 points. The higher the score, the better the self-care ability. Compare the changes of patients' scale scores before and after intervention

SECONDARY OUTCOMES:
Fasting Glucose, Glu | 12months
  Comparison of changes in indicators before and after intervention
Low Density Lipoprotein, LDL | 12 months
  Comparison of changes in indicators before and after intervention
The self rated health status of the patients | 12 months
  Draw a scale with a minimum of 0 and a maximum of 100. 0 represents the worst health condition in the patient's mind, and 100 represents the best health condition in the patient's mind.
  Please mark the health status of the participants on the scale to help them reflect the health status
Total Cholesterol, TC | 12 months
  Comparison of changes in indicators before and after intervention

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Funnell MM, Anderson RM, Arnold MS, Barr PA, Donnelly M, Johnson PD, Taylor-Moon D, White NH. Empowerment: an idea whose time has come in diabetes education. Diabetes Educ. 1991 Jan-Feb;17(1):37-41. doi: 10.1177/014572179101700108. PMID 1986902
- [Result] Wang J, Zhang L, Wang F, Liu L, Wang H; China National Survey of Chronic Kidney Disease Working Group. Prevalence, awareness, treatment, and control of hypertension in China: results from a national survey. Am J Hypertens. 2014 Nov;27(11):1355-61. doi: 10.1093/ajh/hpu053. Epub 2014 Apr 3. PMID 24698853
- [Result] Danaei G, Finucane MM, Lin JK, Singh GM, Paciorek CJ, Cowan MJ, Farzadfar F, Stevens GA, Lim SS, Riley LM, Ezzati M; Global Burden of Metabolic Risk Factors of Chronic Diseases Collaborating Group (Blood Pressure). National, regional, and global trends in systolic blood pressure since 1980: systematic analysis of health examination surveys and epidemiological studies with 786 country-years and 5.4 million participants. Lancet. 2011 Feb 12;377(9765):568-77. doi: 10.1016/S0140-6736(10)62036-3. Epub 2011 Feb 3. PMID 21295844
- [Result] Institute of Medicine (US) Committee on Health Literacy; Nielsen-Bohlman L, Panzer AM, Kindig DA, editors. Health Literacy: A Prescription to End Confusion. Washington (DC): National Academies Press (US); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK216032/ PMID 25009856
- [Result] Sperber NR, Bosworth HB, Coffman CJ, Lindquist JH, Oddone EZ, Weinberger M, Allen KD. Differences in osteoarthritis self-management support intervention outcomes according to race and health literacy. Health Educ Res. 2013 Jun;28(3):502-11. doi: 10.1093/her/cyt043. Epub 2013 Mar 22. PMID 23525779
- [Result] McNaughton CD, Jacobson TA, Kripalani S. Low literacy is associated with uncontrolled blood pressure in primary care patients with hypertension and heart disease. Patient Educ Couns. 2014 Aug;96(2):165-70. doi: 10.1016/j.pec.2014.05.007. Epub 2014 May 14. PMID 24882088
- [Result] Pandit AU, Tang JW, Bailey SC, Davis TC, Bocchini MV, Persell SD, Federman AD, Wolf MS. Education, literacy, and health: Mediating effects on hypertension knowledge and control. Patient Educ Couns. 2009 Jun;75(3):381-5. doi: 10.1016/j.pec.2009.04.006. Epub 2009 May 12. PMID 19442477
- [Result] Morrow D, Clark D, Tu W, Wu J, Weiner M, Steinley D, Murray MD. Correlates of health literacy in patients with chronic heart failure. Gerontologist. 2006 Oct;46(5):669-76. doi: 10.1093/geront/46.5.669. PMID 17050758
- [Result] Shibuya A, Inoue R, Ohkubo T, Takeda Y, Teshima T, Imai Y, Kondo Y. The relation between health literacy, hypertension knowledge, and blood pressure among middle-aged Japanese adults. Blood Press Monit. 2011 Oct;16(5):224-30. doi: 10.1097/MBP.0b013e32834af7ba. PMID 21857504
- [Result] Pleasant A. Advancing health literacy measurement: a pathway to better health and health system performance. J Health Commun. 2014 Dec;19(12):1481-96. doi: 10.1080/10810730.2014.954083. PMID 25491583
- [Result] Chinenye S, Young EE. Diabetes conversation map in Nigeria: A new socioeducational tool in diabetes care. Indian J Endocrinol Metab. 2013 Nov;17(6):1009-11. doi: 10.4103/2230-8210.122613. PMID 24381876
- [Derived] Gan W, Zhang Q, Yang D, Yin J, Wang Y, Song L, Chen T, Qi H. A behavior change wheel-based interactive pictorial health education program for hypertensive patients with low blood pressure health literacy: study protocol for a randomized controlled trial. Trials. 2022 May 3;23(1):369. doi: 10.1186/s13063-022-06300-1. PMID 35505379